# **Statistical Analysis Plan Amendment 1**

**Study ID:** 218350

**Official Title of Study:** A Phase III, open-label, randomized, controlled, multi-country study to evaluate the immune response, safety and reactogenicity of an RSVPreF3 OA investigational vaccine when co-administered with FLU aQIV (inactivated influenza vaccine – adjuvanted) in adults aged 65 years and above.

NCT number: NCT05568797

**Date of Document:** 21 Dec 2022

**Information Type:** Statistical Analysis Plan (SAP)

## TITLE PAGE

**Protocol Title:** A Phase III, open-label, randomized, controlled, multi-

country study to evaluate the immune response, safety and reactogenicity of an RSVPreF3 OA investigational vaccine when co-administered with FLU aQIV (inactivated influenza vaccine – adjuvanted) in adults aged 65 years and above.

Study Number: 218350

**Compound Number:** GSK3844766A

**Abbreviated Title:** RSV OA=ADJ-017

**Sponsor Name:** GlaxoSmithKline Biologicals SA (GSK)

Regulatory Agency

IND 18540 RSV PreF3 Older Adult

Identifier Number(s)

**Registry** ID

Clintrials.gov Not yet available

XBU Statistical Analysis Plan (SAP) Template v2.0 17 January 2022

Copyright 2022 the GlaxoSmithKline group of companies. All rights reserved. Unauthorized copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| TIT | LE PAC | GE | 1 |
| VEI | RSION | HISTORY | 5 |
| 1. | INTRO | DDUCTION | 6 |
| | 1.1.<br>1.2. | | 6 |
| 2. | | ISTICAL HYPOTHESES | |
| | 2.1. | Multiplicity Adjustment | 10 |
| 3. | ANAL | YSIS SETS | |
| | 3.1. | Criteria for eliminating data from Analysis Sets | |
| | | 3.1.1. Elimination from Exposed Set (ES) | |
| | | 3.1.2. Elimination from Per Protocol Set (PPS) | 11 |
| 4. | STAT | ISTICAL ANALYSES | 14 |
| | 4.1. | General Considerations | 14 |
| | | 4.1.1. General Methodology | |
| | | 4.1.2. Definition: | |
| | 4.2. | Primary Endpoints Analyses | |
| | | 4.2.1. Between groups assessment | |
| | | 4.2.2. Main analytical approach | |
| | 4.0 | 4.2.3. Sensitivity analyses | |
| | 4.3. | Secondary Endpoints Analyses | |
| | | 4.3.1. Immunogenicity analysis | |
| | | 4.3.1.1. Between groups assessment | |
| | | 4.3.1.2. Within groups assessment | |
| | 4.4. | | |
| | 4.4. | Exploratory Endpoints Analyses | Z1 |
| | 4.5. | Safety Analyses | |
| | | 4.5.1. COVID-19 Assessment and COVID-19 AEs | |
| | 4.6. | Other Analyses | |
| | 4.7. | Interim Analyses | |
| | 4.8. | Changes to Protocol Defined Analyses | 23 |
| 5. | SAMP | PLE SIZE DETERMINATION | 23 |
| 6. | SLIPP | ORTING DOCUMENTATION | 25 |
| ٥. | 6.1. | Appendix 1 Study Population Analyses | |
| | J | 6.1.1. Participant Disposition | |
| | | 6.1.2. Demographic and Baseline Characteristics | |
| | | 6.1.3. Protocol Deviations | |
| | | 6.1.4. Concomitant Medications | |
| | | 6.1.5. Concomitant Vaccinations | |
| | | 6.1.6. Additional Analyses Due to the COVID-19 Pandemic | 26 |

# **CONFIDENTIAL**

| 6.2. | Appendi | x 2 Data De | erivations Rule | 26 |
|---|---|---|---|---|
| | 6.2.1. | | | |
| | 6.2.2. | | | |
| | | 6.2.2.1. | | |
| | | 6.2.2.2. | | |
| | | 6.2.2.3. | | |
| | 6.2.3. | Data deriv | | |
| | | 6.2.3.1. | | |
| | | 6.2.3.2. | | |
| | | 6.2.3.3. | | |
| | | 6.2.3.4. | Numerical serology results | 29 |
| | | 6.2.3.5. | Geometric mean titers (GMTs) and | |
| | | | | 29 |
| | | 6.2.3.6. | | |
| | | 6.2.3.7. | Duration of events | 30 |
| | | 6.2.3.8. | Counting rules for combining solicited and | |
| | | | unsolicited adverse events | 30 |
| | | 6.2.3.9. | Counting rules for occurrences of solicited | |
| | | | events | 30 |
| | | 6.2.3.10. | Counting rules for occurrence of unsolicited | |
| | | | adverse events | 31 |
| | 6.2.4. | Display of | decimals | 32 |
| | | 6.2.4.1. | Percentages | 32 |
| | | 6.2.4.2. | | |
| | | 6.2.4.3. | Demographic/baseline characteristics statistics | 32 |
| | | 6.2.4.4. | Serological summary statistics | 32 |
| DEEE | DENCES | | | 33 |
| | | 6.2.1.<br>6.2.2.<br>6.2.3. | 6.2.1. Attributing 6.2.2.1. 6.2.2.2. 6.2.2.3. 6.2.3.1. 6.2.3.2. 6.2.3.3. 6.2.3.4. 6.2.3.5. 6.2.3.6. 6.2.3.7. 6.2.3.8. 6.2.3.9. 6.2.3.10. 6.2.4.1. 6.2.4.2. 6.2.4.3. 6.2.4.4. | 6.2.1. Attributing events to vaccine doses. 6.2.2. Handling of missing data 6.2.2.1. Dates 6.2.2.2. Laboratory data 6.2.2.3. Daily recording of solicited events. 6.2.3. Data derivation. 6.2.3.1. Age at first dose in years 6.2.3.2. Age category at vaccination 6.2.3.3. Temperature 6.2.3.4. Numerical serology results 6.2.3.5. Geometric mean titers (GMTs) and concentrations (GMCs) 6.2.3.7. Duration of events 6.2.3.8. Counting rules for combining solicited and unsolicited adverse events. 6.2.3.9. Counting rules for occurrences of solicited events 6.2.3.10. Counting rules for occurrence of unsolicited adverse events |

# CONFIDENTIAL

218350

# **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Populations for analyses | 10 |
| Table 2 | List of elimination codes | 11 |
| Table 3 | Overall power to demonstrate primary objectives: non-inferiority of the immunogenicity of the RSVPreF3 OA investigational vaccine when co-administered with FLU aQIV compared to when administered alone – assuming approximately 462 participants are available in each group | 24 |
| Table 4 | Evaluation of non-inferiority in terms of HI antibody SCR when FLU aQIV is co-administered with the RSVPreF3 OA investigational vaccine compared to FLU aQIV when administered alone assuming approximately 462 participants are available in each group for a range of plausible SCRs | 25 |
| Table 5 | Intensity grading scale for solicited events | 31 |

# **VERSION HISTORY**

| SAP<br>Version | Approval Date | Protocol Version<br>(Date) on which<br>SAP is Based | Change | Rationale |
|---|---|---|---|---|
| SAP | 01 Sep 2022 | 24 March 2022 | Not<br>Applicable | Original version |
| SAP<br>amendment<br>1 | 21 Dec 2022 | Amendment 1: 13<br>December 2022 | Addition of<br>RSV-B as<br>part of<br>primary<br>endpoint | Protocol<br>Amendment<br>1 |

# 1. INTRODUCTION

The purpose of this SAP is to describe the planned analyses to be included in the clinical study report (CSR) for Study RSV OA=ADJ-017 (218350). Details of the planned analysis are provided.

# 1.1. Objectives, Estimands and Endpoints

| Objectives | | | Endpoints and Estimands |
|---|---|---|---|
| | Prin | nary | |
| • | To demonstrate the non-inferiority of the FLU vaccine when co-administered with the RSVPreF3 OA investigational vaccine compared to the FLU vaccine administered alone. | • | HI antibody titers for each of the FLU vaccine strains expressed as group GMT ratio, one month after the FLU vaccine dose. |
| • | To demonstrate the non-inferiority of the RSVPreF3 OA investigational vaccine when co-administered with the FLU vaccine compared to the RSVPreF3 OA investigational vaccine administered alone. | • | RSV-A neutralization antibody titers expressed as group GMT ratio, one month after the RSVPreF3 OA investigational vaccine dose. |
| • | To demonstrate the non-inferiority of the RSVPreF3 OA investigational vaccine when co-administered with the FLU vaccine compared to the RSVPreF3 OA investigational vaccine administered alone. | • | RSV-B neutralization antibody titers expressed as group GMT ratio, one month after the RSVPreF3 OA investigational vaccine dose. |
| | Seco | ndar | у |
| • | To evaluate the non-inferiority of the FLU vaccine when co-administered with the RSVPreF3 OA investigational vaccine compared to the FLU vaccine administered alone. | • | HI seroconversion status for each of the FLU vaccine strains expressed as SCR between groups, one month after the FLU vaccine dose. |
| • | To evaluate the humoral immune response to the RSVPreF3 OA investigational vaccine when co-administered with the FLU vaccine or | • | RSV-A neutralization antibody titers expressed as MGI at one month after the RSVPreF3 OA investigational vaccine dose. |
| | administered alone. | • | RSV-B neutralizing antibody titers expressed as MGI at one month after the RSVPreF3 OA investigational vaccine dose. |
| • | To evaluate the humoral immune response to the FLU vaccine when co-administered with the | • | HI antibody titers for each of the FLU vaccine strains expressed as GMT, at Day 1 and Day 31. |
| | RSVPreF3 OA investigational vaccine or administered alone. | • | HI seroconversion status for each of the FLU vaccine strains expressed as SCR, from Day 1 to Day 31. |
| | | • | HI seroprotection status for each of the FLU vaccine strains expressed as SPR, at Day 1 and Day 31. |
| | | • | HI antibody titers for each of the FLU vaccine strains expressed as MGI, one month after the FLU vaccine dose. |
| • | To evaluate the safety and reactogenicity following administration of the RSVPreF3 OA investigational vaccine and the FLU vaccine, co-administered or administered alone. | • | Percentage of participants reporting each solicited event with onset within 7 days after vaccine administration (i.e., the day of vaccination and 6 subsequent days). |
| | | • | Percentage of participants reporting unsolicited AEs (pIMD, non-serious AE or serious AE) within 30 days after vaccine administration (i.e., the day of vaccination and 29 subsequent days). |

| Objectives | Endpoints and Estimands |
|---|---|
| | Percentage of participants reporting SAEs after vaccine administration (Day 1) up to study end (6 months after last vaccination). |
| | <ul> <li>Percentage of participants reporting pIMDs after<br/>vaccine administration (Day 1) up to study end<br/>(6 months after last vaccination).</li> </ul> |
| CCI | |

FLU vaccine refers to FLU aQIV

**AE** = adverse event; **GCI**; **GMT** = geometric mean titer; **HI** = hemagglutination inhibition; **MGI** = mean geometric increase; **pIMD** = potential immune-mediated disease; **RSVPreF3 OA** = respiratory syncytial virus PreFusion protein 3 older adult; **SAE** = serious adverse event; **SCR** = seroconversion rate; **SPR** = seroprotection rate:

MGI = geometric mean of the within participant ratios of the post-dose titer over the pre-dose titer.

SCR = percentage of vaccinees who have either a HI pre-dose titer < 1:10 and a post-dose titer  $\geq$  1:40 or a pre-dose titer  $\geq$  1:10 and at least a 4-fold increase in post-dose titer.

SPR = percentage of vaccinees with a serum HI titer ≥ 1:40 that usually is accepted as indicating protection.

## **Primary estimand**

The primary clinical question of interest is to show non-inferiority of the RSVPreF3 OA investigational vaccine and the FLU vaccine when co-administered versus separate administration 1 month apart in eligible participants who complied with the study requirements as defined Per Protocol (refer to Section 3 for the definition of the Per Protocol Set [PPS] used for the primary analysis and to Section 4.2.2 for the statistical method).

# 1.2. Study Design



**AE** = adverse event; **N** = number of participants; **pIMD** = potential immune-mediated disease; **RSV** = respiratory syncytial virus; **SAE** = serious adverse event

### **Design Features**

- Type of study: self-contained.
- Experimental design: Phase III, randomized (ratio 1:1), open-label, multi-country study with 2 parallel groups.
- Study groups:
  - Co-Ad (co-administration) group: Participants receiving the RSVPreF3 OA investigational vaccine co-administered with FLU aQIV (referred to as FLU vaccine).
  - Control group: Participants receiving the FLU aQIV (referred to as FLU vaccine) and the RSVPreF3 OA investigational vaccine in a sequential manner.
- **Duration of the study**: ~6 months for participants in Co-Ad group; ~7 months for participants in Control group.
- Primary completion date: Day 61 (1 month after the RSVPreF3 OA investigational vaccine dose in Control group).
- Control: active comparator, i.e., sequential administration of licensed FLU vaccine and RSVPreF3 OA investigational vaccine.
- Blinding: open-label.
- Vaccination schedule:
  - Co-Ad group: Participants will be receiving both the RSVPreF3 OA investigational vaccine and FLU vaccine at Visit 1 (Day 1).
  - Control group: Participants will be receiving the FLU vaccine at Visit 1 (Day 1) and subsequently the RSVPreF3 OA investigational vaccine at Visit 2 (Day 31).

| Overview of Study Design and Key Features | | | | |
|---|---|---|---|---|
| Study intervention | Study Groups | Number of<br>Participants | Age<br>(Min-Max) | Study Interventions |
| | Co-Ad | ~514 | ≥ 65 years | RSVPreF3 OA investigational vaccine |
| | | | • | FLU aQIV |
| | Control | ~514 | ≥ 65 years | RSVPreF3 OA investigational vaccine |
| | older adult | | OA = respiratory | FLU aQIV syncytial virus PreFusion protein 3 |
| Interim Analysis | No interim analysis | s is planned | | |

## 2. STATISTICAL HYPOTHESES

The study includes the following confirmatory primary objectives.

• To demonstrate the non-inferiority of FLU vaccine when co-administered with the RSVPreF3 OA investigational vaccine compared to FLU vaccine administered alone in terms of HI GMT ratio for each of the FLU vaccine strains at 1 month after the FLU vaccine (i.e., at Day 31 [Visit 2] for both groups).

## **Null hypothesis vs. Alternative hypothesis:**

H<sub>0</sub>: 
$$\mu_{\text{Control group}}$$
-  $\mu_{\text{Co-Ad group}} > \log(1.5)$  vs. H<sub>a</sub>:  $\mu_{\text{Control group}}$ - $\mu_{\text{Co-Ad group}} \leq \log(1.5)$ 

where  $\mu$  represents the estimated mean of log transformed HI antibody titers at 1 month after the FLU vaccine dose. The null hypothesis will be rejected if the upper limit of the two-sided 95% CI for the group GMT ratio (Control group divided by Co-Ad group) in HI antibody titers for each of the FLU vaccine strains 1 month after the FLU vaccine  $\leq 1.5$ 

• To demonstrate the non-inferiority of RSVPreF3 OA investigational vaccine when co-administered with the FLU vaccine compared to RSVPreF3 OA investigational vaccine administered alone in terms of RSV-A neutralization antibody GMT ratio at 1 month after the RSVPreF3 OA investigational vaccine dose (i.e., at Day 31 [Visit 2] for the Co-Ad group and at Day 61 [Visit 4] for the Control group).

### **Null hypothesis vs. Alternative hypothesis:**

```
H<sub>0</sub>: \mu_{\text{Control group}} - \mu_{\text{Co-Ad group}} > \log(1.5) vs. H<sub>a</sub>: \mu_{\text{Control group}} - \mu_{\text{Co-Ad group}} \leq \log(1.5)
```

where  $\mu$  represents the estimated mean of log transformed RSV-A neutralization antibody titers at 1 month after the RSVPreF3 OA investigational vaccine dose. The null hypothesis will be rejected if the upper limit of the two-sided 95% confidence interval (CI) for the group GMT ratio (Control group divided by Co-Ad group) in RSV-A neutralization antibody titers 1 month after the RSVPreF3 OA investigational vaccine dose  $\leq$  1.5.

 To demonstrate the non-inferiority of RSVPreF3 OA investigational vaccine when co-administered with the FLU vaccine compared to RSVPreF3 OA investigational vaccine administered alone in terms of RSV-B neutralization antibody GMT ratio at 1 month after the RSVPreF3 OA investigational vaccine dose (i.e., at Day 31 [Visit 2] for the Co-Ad group and at Day 61 [Visit 4] for the Control group).

# **Null hypothesis vs. Alternative hypothesis:**

```
H<sub>0</sub>: \mu_{\text{Control group}} - \mu_{\text{Co-Ad group}} > \log(1.5) vs. H<sub>a</sub>: \mu_{\text{Control group}} - \mu_{\text{Co-Ad group}} \leq \log(1.5)
```

where  $\mu$  represents the estimated mean of log transformed RSV-B neutralization antibody titers at 1 month after the RSVPreF3 OA investigational vaccine dose. The null hypothesis will be rejected if the upper limit of the two-sided 95% confidence interval (CI) for the group GMT ratio (Control group divided by Co-Ad group) in RSV-A neutralization antibody titers 1 month after the RSVPreF3 OA investigational vaccine dose  $\leq 1.5$ .

# 2.1. Multiplicity Adjustment

Using a nominal alpha of 2.5% for each of them will ensure the global type I error for the primary objectives is controlled below 2.5%.

# 3. ANALYSIS SETS

The following analysis sets will be used for this study:

Table 1 Populations for analyses

| Analysis set | Description |
|---|---|
| Enrolled set | Participants who were randomized or received study intervention or have |
| | undergone an invasive procedure. |
| Exposed set | All participants who received a study intervention. Analysis per group is based on the study intervention administered. |
| Per Protocol set | All eligible participants: |
| | <ul> <li>who received at least one study intervention as Per Protocol in the control group and all study interventions in the Co-Ad group,</li> <li>had immunogenicity results pre- and post-dose,</li> </ul> |
| | <ul> <li>complied with blood draw intervals (mentioned below) (contribution of participants to Per Protocol set at specific timepoint will be defined by timepoint),</li> </ul> |
| | without intercurrent medical conditions that may interfere with immunogenicity and, |
| | <ul> <li>without prohibited concomitant medication/vaccination.</li> </ul> |

Intervals for the Co-Ad group: Visit1(D1)-Visit2 (D31) =30-37 days

Intervals for the Control group: Visit1(D1)-Visit2(D31) =30-37 days, Visit2(D31)-Visit3(D45) =12 - 16 days, Visit2(D31)-Visit4(D61) =30-37 days

# 3.1. Criteria for eliminating data from Analysis Sets

Elimination codes will be used to identify participants to be eliminated from analysis. Detail is provided below for each set.

# 3.1.1. Elimination from Exposed Set (ES)

Code 1030 (Study intervention not administered at all), 800 (Fraudulent data) and code 900 (invalid informed consent) will be used for identifying participants eliminated from ES (see Table 2).

# 3.1.2. Elimination from Per Protocol Set (PPS)

A participant will be excluded from the populations for analysis under the following conditions:

- For codes 800, 900, 1030, 1050 and 2020: participants will be eliminated for all visits.
- For codes 1070, 1080, 1090: participants will be eliminated from a specific visit (at which the condition is met) onwards for the specific group/antigens.
- For codes 1040,2010, 2040, 2050, 2080: participants will be eliminated from a specific visit (at which the condition is met) onwards.
- For codes 2090, 2100, 2120: participants will be eliminated at the specific visit at which the condition is met.

#### Table 2 List of elimination codes

| Code | Condition under which the code is used | Visit /Contact(timepoints) where the code is checked | Visit from when it is applicable | Applicable for analysis set/endpoint |
|---|---|---|---|---|
| 800 | Fraudulent data | All | All | ES and PPS<br>for analysis of<br>immunogenicity |
| 900 | Invalid informed consent | All | All | ES and PPS<br>for analysis of<br>immunogenicity |
| 1030 | Study intervention not administered at all | All | All | ES and PPS<br>for analysis of<br>immunogenicity |
| 1040 | Administration of concomitant vaccine(s) forbidden in the protocol Use of any investigational or non- registered vaccine other than the study interventions during the period beginning 30 days before the first dose of study interventions, or planned use during the study period. Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first study intervention administration and ending 30 days after the last study intervention administration. | Visit 1,2 for the Co-ad group. Visit 1,2,3*,4 for the control group | From the specific visit the condition is met | PPS for analysis of immunogenicity |

| Code | Condition under which the code is used | Visit<br>/Contact(timepoints)<br>where the code is<br>checked | Visit from when it is applicable | Applicable for analysis set/endpoint |
|---|---|---|---|---|
| | In the case of COVID-19 vaccines, this time window can be decreased to 14 days before and after each study intervention administration provided this COVID-19 vaccine use is in line with local governmental recommendations. Note: In case an emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) is recommended and/or organized by the public health authorities, outside the routine immunization program, the time period described above can be reduced if necessary for that vaccine provided it is used according to the local governmental recommendations and that the Sponsor is notified accordingly. | | | |
| 1050 | Randomization failure: Participant not randomized in the correct group (To be attributed by Statistician only; Check SBIR, replacement, vaccine administration) | Visit 1 | All | PPS for<br>analysis of<br>immunogenicity |
| 1070 | Vaccine administration not according to protocol Incomplete vaccination course Participant was vaccinated with the correct vaccine but containing a lower volume Wrong replacement or study vaccine administered (not compatible with the vaccine regimen associated to the treatment number) Route of the study vaccine is not intramuscular Side of administration wrong (for Co-ad group if both vaccines are given in the same arm) Wrong reconstitution of administered vaccine | Vaccination visit(s) 1 or 1 and 2 as applicable | From the specific visit (1 or 2) the condition is met as applicable for the respective group/antigen | PPS for analysis of immunogenicity |
| 1080 | Vaccine temperature deviation Vaccine administered despite a GMP nogo temperature deviation | Vaccination visit(s) 1 or 1 and 2 as applicable | From the specific visit (1 or 2) the condition is met as applicable for the respective group/antigen | PPS for<br>analysis of<br>immunogenicity |
| 1090 | Expired vaccine administered | Vaccination visit(s) 1<br>or 1 and 2 as<br>applicable | From the specific visit (1 or 2) the condition is met as applicable for the respective group/antigen | PPS for<br>analysis of<br>immunogenicity |
| 2010 | Protocol violation linked to inclusion/exclusion criteria | Visit 1,2 for the Co-ad group. | From the specific visit (1,2,3* or 4) | PPS for analysis of immunogenicity |

| Code | Condition under which the code is used | Visit<br>/Contact(timepoints)<br>where the code is<br>checked | Visit from when it is applicable | Applicable for analysis set/endpoint |
|---|---|---|---|---|
| | All inclusion/exclusion criteria defined in the protocol to be checked. | Visit 1,2,3*,4 for the control group | the condition is met. | |
| 2020 | All Pre-dose results are missing:<br>RSV-A, RSV-B and HI for the FLU vaccine<br>strains | Co-Ad group: Visit 1<br>Control group: Visit 1<br>and Visit 2 | All | PPS for analysis of immunogenicity |
| 2040 | Administration of any medication forbidden by the protocol Use of any investigational or non-registered product (drug or medical device) other than the study interventions during the period beginning 30 days before the first dose of study interventions, or planned use during the study period. Administration of long-acting immune-modifying drugs or planned administration at any time during the study period (e.g., infliximab). Administration of immunoglobulins and/or any blood products or plasma derivatives planned administration during the study period. Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs planned administration during the study period. For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent. Inhaled and topical steroids are allowed. | Visit 1,2 for the Co-ad group. Visit 1,2,3*,4 for the control group | From the specific visit (1,2,3* or 4) the condition is met | PPS for analysis of immunogenicity |
| 2050 | Intercurrent medical condition: Participants may be eliminated from the PPS for immunogenicity if, during the study, they incur a condition that has the capability of altering their immune response (intercurrent medical condition) or are confirmed to have an alteration of their initial immune status. | Visit 1,2 for the Co-ad group. Visit 1,2,3*,4 for the control group | From the specific visit (1,2,3* or 4) the condition is met | PPS for<br>analysis of<br>immunogenicity |
| 2080 | Participants did not comply with vaccination schedule for the control group number of days between dose 1 and dose 2 is outside [30-37 days] | Visit 2 | Visit 3 for the control group | PPS for analysis of immunogenicity |
| 2090 | Participants did not comply with blood sample schedule: Co-Ad group: Number of days between vaccination (visit1) and blood sample (visit2) is outside [30-37] days Control group: Number of days between vaccination (visit1) and blood sample (visit2) or (visit2) and blood sample (visit4) is outside [30-37] days Or | Visit 2, Visit 3*, Visit 4 as applicable for the group | At the specific visit (2,3* or 4) the condition is met as applicable for the respective group | PPS for<br>analysis of<br>immunogenicity |

| Code | Condition under which the code is used | Visit /Contact(timepoints) where the code is checked | Visit from when it is applicable | Applicable for analysis set/endpoint |
|---|---|---|---|---|
| | blood sample (visit2) and blood sample (visit3) are outside [12-16] days | | | |
| 2100 | Serological results not available at the post-dose time point for all antigens tested at that particular time point. | Visit 2,3*,4 | At the specific visit (2,3* or 4) the condition is met as applicable for the respective group | PPS for<br>analysis of<br>immunogenicity |
| 2120 | Obvious incoherence/abnormality or error in laboratory data Unreliable released data as a result of confirmed sample mismatch or confirmed inappropriate sample handling at lab | Visit 2, Visit 3 | At the specific visit (2,3* or 4) the condition is met as applicable for the respective group | PPS for<br>analysis of<br>immunogenicity |

**ES** = exposed set; **GMP** = Good Manufacturing Practices; **HI** = hemagglutination inhibition; **PPS** = Per Protocol set

# 4. STATISTICAL ANALYSES

## 4.1. General Considerations

# 4.1.1. General Methodology

95% CI for proportion will be based on exact Clopper-Pearson CI [Clopper, 1934].

95% CI for group difference in proportion will be based on Miettinen and Nurminen CI [Miettinen, 1985].

The group adjusted GMT ratio will be based on a back transformation of group contrast in an ANCOVA model applied to the logarithm-transformed titers.

<u>Primary Analysis</u>: The ANCOVA model will include the treatment group and age category (age at vaccination: 65-69, 70-79 or ≥80 years) as fixed effects and the pre-dose log-10 titer as regressors.

<u>Sensitivity Analysis</u>: The ANCOVA model will include the treatment group and age category (age at vaccination: 65-69, 70-79 or ≥80 years) as fixed effects, center as the random effect and the pre-dose log-10 titer as regressors.

95% CI for GMT and GMT ratio will be based on a back transformation of student CI for the mean and difference of means (for GMT ratio) respectively of log-transformation (i.e., 10^CI).

#### 4.1.2. Definition:

### • For all endpoints:

The baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

MGI (mean geometric increase): The geometric mean of the within participant ratios of the post-dose titer over the pre-dose titer.

## • For the RSV antigens:

A seronegative participant will be defined as a participant whose antibody titer/concentration is below the cut-off value of the assay. A seropositive participant is a participant whose antibody titer/concentration is greater than or equal to the cut-off value of the assay.

# • For the FLU antigens:

SCR (seroconversion rate): The percentage of vaccinees who have either a HI predose titer < 1:10 and a post-dose titer  $\ge 1:40$  or a pre-dose titer  $\ge 1:10$  and at least a four-fold increase in post-dose titer.

HI SPR (seroprotection rate): The percentage of vaccinees with a serum HI titer  $\geq 1:40$  that usually is accepted as indicating protection.

# 4.2. Primary Endpoints Analyses

The primary analysis will be based on the PPS for analysis of immunogenicity. If, in any vaccine group, the percentage of vaccinated participants with serological results excluded from the PPS for analysis of immunogenicity is 5% or more, a second analysis based on the ES will be performed to complement the PPS analysis.

# 4.2.1. Between groups assessment

- The 2-sided 95% CI for the group GMT ratio in terms of HI antibody titers for each of the FLU vaccine strains between RSVPreF3 OA investigational vaccine administered alone (Control group) over RSVPreF3 OA investigational vaccine when co-administered with the FLU vaccine (Co-Ad group) will be computed at 1 month after the FLU vaccine (i.e., at Day 31 [Visit 2] for both groups).
- The 2-sided 95% CI for the group GMT ratio in terms of RSV-A neutralizing antibody titers between RSVPreF3 OA investigational vaccine administered alone (Control group) over RSVPreF3 OA investigational vaccine when co-administered with the FLU vaccine (Co-Ad group) will be computed at 1 month after the RSVPreF3 OA investigational vaccine dose (i.e., at Day 31 [Visit 2] for the Co-Ad group and at Day 61 [Visit 4] for the Control group).
- The 2-sided 95% CI for the group GMT ratio in terms of RSV-B neutralizing antibody titers between RSVPreF3 OA investigational vaccine administered alone (Control group) over RSVPreF3 OA investigational vaccine when co-administered with the FLU vaccine (Co-Ad group) will be computed at 1 month after the

RSVPreF3 OA investigational vaccine dose (i.e., at Day 31 [Visit 2] for the Co-Ad group and at Day 61 [Visit 4] for the Control group).

The results will be presented in tables as well as graphs using forest plots.

## 4.2.2. Main analytical approach

The 2-sided 95% CI for group adjusted GMT ratio will be derived from **an ANCOVA model** on **log**<sub>10</sub> transformed titer. The model will include the treatment group and age category (age at vaccination: 65-69, 70-79 or ≥80 years) as fixed effects, and the pre-dose log10-transformed titer as covariate. Missing data will not be replaced. Titers below the assay cut-off will be replaced by half the assay cut-off, titers above the upper limit of quantification (ULOQ) will be replaced by the ULOQ.

Success criteria for non-inferiority and testing sequence:

The following testing sequence will be used:

1<sup>st</sup> sequence:

• The upper limit of the 2-sided 95% CI of the GMT ratio (Control group divided by Co-Ad group) for each of the FLU vaccine strains are ≤1.5.

#### **AND**

• The upper limit of the 2-sided 95% CI of the GMT ratio (Control group divided by Co-Ad group) for RSV-A neutralization antibodies is ≤1.5.

2<sup>nd</sup> sequence:

• The upper limit of the 2-sided 95% CI of the GMT ratio (Control group divided by Co-Ad group) for RSV-B neutralization antibodies is ≤1.5.

Testing will progress in the 2<sup>nd</sup> sequence only if the 1st sequence is a success, so that no further adjustment of alpha is required.

Here is an example of SAS code that will be used:

```
proc mixed data=data_in;
class agecat trt_grp;
model log10(titer day x) = log10(pre_dose) agecat trt_grp;
lsmeans trt_grp/cl pdiff alpha=0.05;
run;
```

# 4.2.3. Sensitivity analyses

As for the main analytical approach an ANCOVA model will be performed with the treatment group and age category (age at vaccination: 65-69, 70-79 or ≥80 years) as fixed effects, **center as random effect** and the pre-dose log10-transformed titer as covariate.

In case the model with random effect does not converge we proceed with center as a fixed effect.

Here is an example of SAS code that will be used:

```
proc mixed data=data_in;
class agecat trt_grp center;
model log10(titer day x) = log10(pre_dose) agecat trt_grp;
random intercept/subject=center;
lsmeans trt_grp/cl pdiff alpha=0.05;
run;
```

# 4.3. Secondary Endpoints Analyses

# 4.3.1. Immunogenicity analysis

The primary analysis of secondary immunogenicity endpoints will be based on the PPS for analysis of immunogenicity. If, in any vaccine group, the percentage of vaccinated participants with serological results excluded from the PPS for analysis of immunogenicity is 5% or more, a second analysis based on the ES will be performed to complement the PPS analysis.

## 4.3.1.1. Between groups assessment

• The asymptotic standardized 95% CI for the difference in seroconversion rate (Control group minus Co-Ad group) will be computed at 1 month after the FLU vaccine (i.e., at Day 31 [Visit 2] for both groups).

Reference criteria for evaluation of non-inferiority:

The upper limit of the 2-sided 95% CI on the group difference (Control group minus Co-Ad group) in seroconversion rate is  $\leq$ 10% for anti-HI antibodies.

All between groups analyses of secondary endpoints presented in this section will be descriptive with the aim to characterize the difference in immunogenicity between groups. These descriptive analyses should be interpreted with caution considering that there is no adjustment for multiplicity for these comparisons.

# 4.3.1.2. Within groups assessment

For each group, at each time point that blood samples are collected (except Day 45) for humoral immune response and for each assay (unless otherwise specified):

- Percentage of participants above pre-defined assay cut-off and their exact 95% CI will be tabulated.
- Percentage of participants above seroprotection/seroconversion rate for HI antibody titer and their exact 95% CI will be tabulated.

- GMCs/GMTs and their 95% CI over time will be tabulated and presented graphically (in log10 scale).
- MGI will be tabulated with 95% CI.
- Antibody titer/concentration will be displayed using reverse cumulative curves (both groups and available timepoints (except Day 45) will be presented in the same graph).

The above mentioned descriptive within group immunogenicity analysis will also be generated by age at first vaccination (65-69 YOA, 70-79 YOA, ≥ 70 YOA and ≥80 YOA years).

 Additionally, the CBER and CHMP criteria for HI SPR and SCR will be assessed as follows:

CBER criteria to be evaluated:

- The lower limit (LL) of the 95% CI for SCR should be ≥30% in participants ≥65 YOA.
- The LL of the 95% CI for SPR should be  $\geq$ 60% in participants  $\geq$ 65 YOA.

CHMP criteria to be evaluated:

- At least one of the 3 following criteria should be met:
- the point estimates of SPR >60%, SCR >30%, and MGI >2.0 for elderly > 60 YOA for each of the antigen strains.

These above defined analyses evaluating the CBER and CHMP criteria should be interpreted with caution considering that there is no adjustment for multiplicity for these comparisons.

## 4.3.2. Safety analysis

The safety analysis will be performed on the ES as follows:

• The number and percentage of participants and doses with at least one administration site event AE (solicited and unsolicited), with at least one systemic AE (solicited and unsolicited) and with any AE during the 7-day (i.e., the day of vaccination and 6 subsequent days) and 30-day (i.e., the day of vaccination and 29 subsequent days) follow-up period will be tabulated with exact 95% CI after each dose and overall. The same computations will be done for Grade 3 AEs, for Grade 3 non-serious AEs and for AEs resulting in a medically attended visit.

These analyses will present all solicited and unsolicited AEs, including SAEs and pIMDs (unless otherwise specified).

The above analysis will also be performed for the solicited symptoms only during the 7-day (i.e., the day of vaccination and 6 subsequent days) follow-up period.

• The number and percentage of participants reporting each individual solicited administration site AE (any grade, Grade 3 and resulting in medically attended visit) and solicited systemic AE (any grade, Grade 3 and resulting in medically attended

visit) during the 7-day follow-up period (i.e., the day of vaccination and 6 subsequent days) will be tabulated for each group after each dose and overall. The percentage of doses followed by each individual solicited administration site AE (any grade, Grade 3 and resulting in medically attended visit) and solicited systemic AE (any grade, Grade 3 and resulting in medically attended visit) during the 7-day follow-up period (i.e., the day of vaccination and 6 subsequent days) will be tabulated, with exact 95% CI.

- For fever, the number and percentage of participants reporting fever by half degree (°C) cumulative increments during the 7-day follow-up period (i.e., the day of vaccination and 6 subsequent days) will be tabulated for each group after each dose and overall.
- The percentage of participants with each solicited administration site event and solicited systemic event (any grade and Grade 3) will be represented graphically for each group after each dose.
- The number of days with solicited events reported during the 7-day follow-up period (i.e., the day of vaccination and 6 subsequent days) will be tabulated for each individual solicited event using descriptive statistics (mean, minimum, Q1, median, Q3, maximum). The same computations will be done for Grade 3 solicited events.
- The number of days with solicited events ongoing beyond the 7-day follow-up period (i.e., the day of vaccination and 6 subsequent days) will be tabulated for each individual solicited event using descriptive statistics (mean, minimum, Q1, median, Q3, maximum). The same computations will be done for Grade 3 solicited events.
  - All Analyses described above for solicited AEs will be also generated during only the 4-day follow-up period (i.e., the day of vaccination and 3 subsequent days).
- The number and percentage of participants with any unsolicited AEs during the 30-day follow-up period (i.e., the day of vaccination and 29 subsequent days) with its exact 95% CI will be tabulated by group and by Medical Dictionary for Regulatory Activities (MedDRA) System Organ Class (SOC), High Level Term (HLT) and Preferred Term (PT). Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended visit. The verbatim reports of unsolicited AEs will be reviewed by a physician and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. Every verbatim term will be matched with the appropriate Preferred Term. The above analysis by dose will also be performed.

These analyses will present all unsolicited AEs, including SAEs and pIMDs (unless otherwise specified).

- The number and percentage of participants with at least one report of SAE classified by the MedDRA Primary SOC, HLT and PTs and reported after vaccine administration (Day 1) up to study end (6 months after last vaccination) will be tabulated with exact 95% CI.
- The number and percentage of participants with at least one report of causally related SAE classified by the MedDRA Primary SOC, HLT and PTs and reported after

vaccine administration (Day 1) up to study end (6 months after last vaccination) will be tabulated with exact 95% CI.

- The same tabulation will be presented for fatal SAEs.
- All SAEs will also be described in detail in a tabular listing.
- All pIMDs will also be described in detail in a tabular listing.
- All AEs/SAEs leading to study/intervention discontinuation from dose 1 up to study end will be tabulated.
- The percentage of participants with at least one report of pIMD classified by the MedDRA SOC, HLT and Preferred Terms and reported after vaccine administration (Day 1) up to study end (6 months after last vaccination) will be tabulated with exact 95% CI. The percentage of participants with at least one report of related pIMD classified by the MedDRA SOC, HLT and Preferred Terms and reported after vaccine administration (Day 1) up to study end (6 months after last vaccination) will be tabulated with exact 95% CI.
- For analysis of SAEs/pIMDs from first vaccination up to 6 months **post-last** vaccination, the reporting period will start at vaccination and will end at Day 183 post-last vaccination (i.e., day of last vaccination+183), computed as 6 x 30.5 days=183 days.
- The number and percentage of participants using concomitant medication (any medication and any antipyretic) during the 7-day and the 30-day follow-up period after each dose and overall will be tabulated with exact 95% CI.
- The number and percentage of participants using concomitant vaccination during the 30-day follow-up period after each dose and overall will be tabulated with exact 95% CI.
- Compliance in completing solicited events information will be tabulated after each dose and overall.

Some of the key safety analysis will be generated by age group at first vaccination (65-69 YOA, 70-79 YOA, ≥ 70 YOA and≥80 YOA years) as mentioned below.

- The number and percentage of participants reporting each individual solicited administration site AE (any grade, Grade 3 and resulting in medically attended visit) and solicited systemic AE (any grade, Grade 3 and resulting in medically attended visit) during the 7-day follow-up period (i.e., the day of vaccination and 6 subsequent days) will be tabulated for each group after each dose and overall.
  - The number and percentage of participants with any unsolicited AEs during the 30-day follow-up period (i.e., the day of vaccination and 29 subsequent days) with its exact 95% CI will be tabulated by group and by MedDRA Primary SOC, HLT and PTs
- For clinicaltrials.gov and EudraCT posting purposes, percentage of participants of combined solicited and unsolicited non-serious adverse events during the 30-day follow-up period (i.e., the day of vaccination and 29 subsequent days) will be

produced by System Organ Class and preferred terms and according to occurrence of each event.









Safety analyses are described in Section 4.3.2.

### 4.5.1. COVID-19 Assessment and COVID-19 AEs

Based on the study requirement, related analysis or a listing might be produced for the study if applicable.

A standardized MedDRA Query (SMQ) will be used to identify all COVID-19 AEs.

The overall incidence of COVID-19 AEs and SAEs, COVID-19 AEs leading to study intervention discontinuation, COVID-19 AEs leading to study withdrawal, and severe COVID-19 AEs will be summarized. The incidence of these events at individual PT level can be obtained from the standard AE/SAE summaries.

COVID-19 assessments (confirmed, probable and suspected diagnosis) for participants with COVID-19 AEs will be summarized.

The number and percentage of participants with concomitant vaccination (COVID-19) before and during the study will be tabulated with exact 95% CI.

# 4.6. Other Analyses

Not applicable.

# 4.7. Interim Analyses

No interim analyses are planned for this study.

# 4.8. Changes to Protocol Defined Analyses

No changes from the protocol defined analyses.

# 5. SAMPLE SIZE DETERMINATION

The **target enrollment** will be **1028 participants** (514 in the group receiving the RSVPreF3 OA investigational vaccine co-administered with FLU aQIV [Co-Ad group] and 514 in the Control group where RSVPreF3 OA investigational vaccine and FLU aQIV are administered in a sequential manner). This allows to obtain at least 924 **evaluable participants** (462 in the Co-Ad group and 462 in the Control group) for the

evaluation of the primary objectives, assuming that 10% of the enrolled participants will not be evaluable.

# Participants who withdraw from the study will not be replaced.

Each objective will be evaluated with a nominal type I error of 2.5%.

Table 3 Overall power to demonstrate primary objectives: non-inferiority of the immunogenicity of the RSVPreF3 OA investigational vaccine when co-administered with FLU aQIV compared to when administered alone – assuming approximately 462 participants are available in each group

| Endpoint | Standard<br>deviation of log <sub>10</sub><br>concentration | Reference ratio | Non<br>inferiority<br>margin | Type II<br>error | Power |
|---|---|---|---|---|---|
| FLU non-inferiority* (1-sided to | est with alpha=2.5%) | | | | |
| GMTs HI H1N1 strain | 0.6 | 1.05 | 1.5 | 2.5% | 97.5% |
| GMTs HI H3N2 strain | 0.6 | 1.05 | 1.5 | 2.5% | 97.5% |
| GMTs HI B/Yamagata | 0.6 | 1.05 | 1.5 | 2.5% | 97.5% |
| GMTs HI B/Victoria strain | 0.6 | 1.05 | 1.5 | 2.5% | 97.5% |
| RSV non-inferiority* (1-sided t | est with alpha = 2.5%) | | | | |
| GMTs RSV-A neutralization antibody | 0.45 | 1.05 | 1.5 | 0.1% | 99.9% |
| RSV non-inferiority* (1-sided t | est with alpha = 2.5%) | | | | |
| GMTs RSV-B neutralization | 0.45 | 1.05 | 1.5 | 0.1% | 99.9% |
| antibody | | | | | |
| Global Type II error to show non-inferiority ~10.0% | | | | | |
| Global power | | | | ~90.0% | |

**GMT** = geometric mean titer; **HI** = hemagglutination inhibition; **RSV** = respiratory syncytial virus

\*Pass 2019 alpha = 2.5%, Two-Sample T-Tests for Non-Inferiority Assuming Equal Variance and Equal mean For RSV: non-inferiority limit = 0.176 (=log10[1.5]).

For each FLU vaccine strain: non-inferiority limit = 0.176 (=log10[1.5]).

Reference Ratio= 0.0212 (=log10[1.05])

Considering a potential slight interference of 1.05 in true GMTs in both groups with a common population standard error of 0.45 for the RSV-A and RSV-B neutralization antibodies and 0.6 for each of the FLU strains in log<sub>10</sub> transformed concentration, the study has at least 90.0% power to meet the primary objectives.

### Nominal powers to evaluate the secondary objective

The nominal power to evaluate the non-inferiority on SCR for each of the FLU strains is above 86%, depending on the plausible rates.

Table 4 Evaluation of non-inferiority in terms of HI antibody SCR when FLU aQIV is co-administered with the RSVPreF3 OA investigational vaccine compared to FLU aQIV when administered alone assuming approximately 462 participants are available in each group for a range of plausible SCRs

| N evaluable<br>participants per<br>group | Threshold | Plausible<br>rates in<br>Control<br>group** | Type II error | Nominal Power |
|---|---|---|---|---|
| | | FLU vaccine: Non-inferiority* in terms of SCR | | |
| 462 | 10% | 70% | 8.7% | 91.3% |
| 462 | 10% | 50% | 13.9% | 86.1% |
| 462 | 10% | 35% | 11.0% | 89.0% |
| 462 | 10% | 25% | 6.1% | 93.9% |

**SCR** = Seroconversion Rate.

## 6. SUPPORTING DOCUMENTATION

# 6.1. Appendix 1 Study Population Analyses

A summary of the number of participants in each of the participant level analysis set will be provided.

In this multicentre global study, enrollment will be presented by country.

## 6.1.1. Participant Disposition

The number of participants who withdraw from the study will be tabulated by group according to the reason for drop-out. This analysis will be based on the ES and the PPS.

# 6.1.2. Demographic and Baseline Characteristics

The median, mean, range and standard deviation of age (in years) at first vaccination will be computed by group. The center distribution, distribution of participants in each age category (65-69 YOA, 70-79 YOA, ≥70 YOA and ≥80 YOA) geographical ancestry and sex composition will be presented. This analysis will be based on the ES, the PPS and on the

The number and percentages of participants with medical history classified by the MedDRA Primary SOC, HLT and PTs will be tabulated by group for the ES.

### 6.1.3. Protocol Deviations

The number of participants enrolled into the study as well as the number of participants excluded from per protocol set (PPS) analyses will be tabulated for the total population. This analysis, also broken down by study group, will be based on the ES.

<sup>\*</sup>Pass 2019 alpha = 2.5%, for SCR – Non-inferiority: Proportions – Two independent Proportions – Non-Inferiority Tests for the Difference Between Two Proportions.

<sup>\*\*</sup> SCR observed in the Control group in Zoster-004 study range from 35.3% to 60.9%.

The number of participants enrolled into the study as well as the number of participants excluded from per the ES will be tabulated for the total population. This will be based on all enrolled participants.

#### 6.1.4. Concomitant Medications

The number and percentage of participants and doses using concomitant medication (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) during the 7-day follow-up period (i.e., on the day of vaccination and 6 subsequent days) and during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) will be summarized by group after each vaccine dose and overall.

### 6.1.5. Concomitant Vaccinations

The number and percentage of participants and doses with concomitant vaccination during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) will be summarized by group after each vaccine dose and overall.

# 6.1.6. Additional Analyses Due to the COVID-19 Pandemic

Depending on how the Covid-19 situation evolves, the SAP might be amended to reflect the analysis corresponding to Covid-19.

# 6.2. Appendix 2 Data Derivations Rule

This section contains standard rules for data display and derivation for clinical and epidemiological studies.

# 6.2.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a participant prior to the start of a given event. For example, if the start date of an AE is between Dose 1 and Dose 2, the relative dose will be Dose 1.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the case report form (CRF) using the contents of the flag indicating if the event occurred before or after study dose. If 'after study dose' is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before study dose' is selected, the relative dose for the event will be the dose prior to this one.

# 6.2.2. Handling of missing data

## 6.2.2.1. Dates

When partially completed dates (i.e., dates missing a day and/or month) are used in calculations, the following standard rules will be applied:

• A missing day will be replaced by 15

• A missing day and month will be replaced by June 30<sup>th</sup>.

The following exceptions apply:

When partially completed dates (i.e., with missing day or month) are used in calculations, the following rules will be applied:

- AE start dates with missing day:
  - If the month is not the same as the vaccine dose, then the imputed start date will be the 1<sup>st</sup> of the month.
  - If the event starts in the same month as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the vaccine dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the vaccine dose given during that month.
- AE start dates with missing day and month:
  - If the year is not the same as the vaccine dose, then the imputed start date will be the 1<sup>st</sup> of January.
  - If the event starts in the same year as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first vaccine dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first vaccine dose given during that year.
- AE end dates with missing day: the imputed end date will be the last day of the month (30 or 31) or the study conclusion date whichever comes first.
- AE end dates with missing day and month: the imputed end date will be the last day of the year (31st of December) or the study conclusion date whichever comes first.

All incomplete concomitant medication/vaccination start/end date will follow the rules above.

## 6.2.2.2. Laboratory data

Missing laboratory results (including immunological data) will not be replaced.

### 6.2.2.3. Daily recording of solicited events

An eDiary will be used in this study to capture solicited administration site or systemic events, the following rules are applicable for all solicited events except fever:

• Denominators for the summary of administration site (or systemic) solicited events will be calculated using the number of participants who respond to one of the three questions below:

- The question concerning the occurrence for the **Redness and Swelling** symptoms (i.e., is there any Swelling/Redness at the administration site?).
- The question related to the intensity (i.e.,: Please indicate the intensity of the <symptom>)
- The question related to medically attention (i.e.,: Was advice taken for a healthcare professional for this event?).

For the **Redness and Swelling** symptoms the following rules will also be applied:

- When a participant answer "No" to the question: is there any Swelling/Redness at the administration site? the daily measurements will be imputed as None.
- When a participant answer "Yes" to the question: is there any Swelling/Redness at the administration site? any missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the solicited event summary tables.

The following table shows how participants contribute to each category for a specific solicited event over the Day X to Day Y post-dose period:

| Solicited event category | Participants included in the calculation of the numerator |
|---|---|
| Any | All participants with at least one occurrence of the adverse event at Grade 1, Grade 2, or Grade 3 between Day X and Day Y or with the adverse event marked as present and at least one missing daily recording between Day X and Day Y |
| At least Grade 1 | All participants with at least one occurrence of the adverse event at Grade 1, Grade 2, or Grade 3 between Day X and Day Y |
| At least Grade 2 | All participants with at least one occurrence of the adverse event at Grade 2 or Grade 3 between Day X and Day Y |
| At least Grade 3 | All participants with at least one occurrence of the adverse event at Grade 3 between Day X and Day Y |

For fever, the summary tables will not include the row 'Any'. The missing daily records do not contribute to the number participants reporting fever by half degree (°C):  $\geq 38$ ;  $\geq 38.5, \geq 39, \geq 39.5$  and  $\geq 40$ .

#### 6.2.3. Data derivation

# 6.2.3.1. Age at first dose in years

Age will be calculated as the number of years between the year of birth and the year of first vaccination.

## 6.2.3.2. Age category at vaccination

As only the year of birth will be collected in the eCRF, there might be some discrepancies between the age computed using standard derivation rules and the age category used in SBIR for the minimization.

Therefore, for the analysis by age, the age categories will be determined according to the information entered in SBIR (add name of variable in SDTM), except for "≥65 YOA" category which will be obtained using the derived age because this category is not used in SBIR for minimization.

# 6.2.3.3. Temperature

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

Temperature (Celsius) = ([Temperature (Fahrenheit) - 32] × 5)/9

## 6.2.3.4. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For all the assays available for the study, the following derivation rules apply:

| IS.ISORRES | Derived value |
|----------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is ≤ assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is ≥ assay cut-off | value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is ≥ cut-off | Value |
| "value" and value is > ULOQ | ULOQ |
| All other cases | missing |

Note: The Reverse Cumulative Distribution curves (RCC) generated will not use the ULOQ values but the exact value if the exact value is greater than ULOQ.

### 6.2.3.5. Geometric mean titers (GMTs) and concentrations (GMCs)

GMT or GMC calculations are performed by taking the inverse logarithm of the mean of the log titer or concentration transformations. Non quantifiable antibody titers or concentrations will be converted as described in Section 6.2.3.4 for the purpose of GMT/GMC calculation. Cut-off values are defined by the laboratory before the analysis.

## 6.2.3.6. Onset day

The onset day for an event (e.g., AE, concomitant medication/vaccination) is the number of days between the last study dose and the start date of the event. This is 1 for an event occurring on the same day as a study dose (and reported as starting after study dose).

#### 6.2.3.7. Duration of events

## For the duration of solicited AEs:

• The duration of the event will be calculated as the sum of the individual days with the event reported as Grade 1 or higher or reported as missing during the solicited event period (see Section 6.2.2.3 for missing data). For Grade 3, the duration will be calculated as the sum of individual days with the event reported as Grade 3 or reported as missing during the solicited event period.

# 6.2.3.8. Counting rules for combining solicited and unsolicited adverse events

For output combining solicited and unsolicited adverse events, all serious adverse events will be considered systemic events since the administration site flag is not included in the expedited adverse event CRF pages. Unsolicited adverse events with missing administration site flag will also be considered systemic.

Solicited events will be coded by MedDRA as per the following codes:

| Solicited event | Lower level term code | Corresponding Lower level term decode |
|---|---|---|
| Pain | 10022086 | Injection site pain |
| Erythema | 10022061 | Injection site erythema |
| Swelling | 10053425 | Injection site swelling |
| Fever | 10016558 | Fever |
| Headache | 10019211 | Headache |
| Fatigue | 10016256 | Fatigue |
| Myalgia | 10028411 | Myalgia |
| Arthralgia | 10003239 | Arthralgia |

The latest available MedDRA version will be used for coding

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

### 6.2.3.9. Counting rules for occurrences of solicited events

When the occurrences of solicited events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs. Also, in the case of co-administered study interventions, an administration site event recorded for a participant following multiple study interventions will be counted as only one occurrence.

 Table 5
 Intensity grading scale for solicited events

| Event | Intensity Grade | Parameter |
|---|---|---|
| Pain at administration site 0 | | None |
| | 1 | Mild: Any pain neither interfering with nor preventing normal |
| | | everyday activities. |
| | 2 | Moderate: Painful when limb is moved and interferes with everyday |
| | | activities. |
| | 3 | Severe: Significant pain at rest. Prevents normal everyday activities. |
| Erythema at administration site | | Greatest surface diameter in mm |
| Swelling at administration site | | Greatest surface diameter in mm |
| Temperature* | | Temperature in °C. |
| Headache | 0 | None |
| | 1 | Mild: Headache that is easily tolerated |
| | 2 | Moderate: Headache that interferes with normal activity |
| | 3 | Severe: Headache that prevents normal activity |
| Fatigue 0 | | None |
| | 1 | Mild: Fatigue that is easily tolerated |
| 2 | | Moderate: Fatigue that interferes with normal activity |
| | 3 | Severe: Fatigue that prevents normal activity |
| Myalgia 0 | | None |
| | 1 | Mild: Myalgia that is easily tolerated |
| | 2 | Moderate: Myalgia that interferes with normal activity |
| | 3 | Severe: Myalgia that prevents normal activity |
| Arthralgia | 0 | None |
| | 1 | Mild: Arthralgia that is easily tolerated |
| | 2 | Moderate: Arthralgia that interferes with normal activity |
| | 3 | Severe: Arthralgia that prevents normal activity |

The route for measuring temperature can be oral or axillary. Fever is defined as temperature ≥38.0°C regardless of the location of measurement.

The maximum intensity of local injection site erythema/swelling, and fever will be scored at GSK as follows:

| | Erythema/swelling | Fever |
|----|-------------------|-------------------|
| 0: | ≤20mm | < 38.0°C |
| 1: | >20 - ≤50mm | ≥38.0°C - ≤38.5°C |
| 2: | > 50 - ≤100mm | >38.5°C - ≤39.0°C |
| 3: | >100mm | >39.0°C |

## 6.2.3.10. Counting rules for occurrence of unsolicited adverse events

Unsolicited AE summaries will include SAEs and pIMDs unless specified otherwise.

As per CDISC Vaccines Therapeutic Area guide, the solicited events which continue beyond the observation period are stored in the Adverse Events (AE) domain but will not contribute to the summaries of unsolicited AEs.

Missing severity, relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' when displayed in a statistical output.

# 6.2.4. Display of decimals

# 6.2.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with one decimal except for 100% in which case no decimal will be displayed.

# 6.2.4.2. Differences in percentages

Differences in percentages and their corresponding confidence limits will be displayed with 2 decimals.

### 6.2.4.3. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics (age at first vaccination) will be presented with one decimal.

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maximum and minimum of transformed body temperatures will be displayed with one decimal.

# 6.2.4.4. Serological summary statistics

For each assay, GMT or GMC and their confidence limits will be presented with one decimal, as well as GMT/GMC fold increase from pre-dose.

GMT or GMC group ratios and their confidence limits will be displayed with 2 decimals regardless of the actual values.

# 7. REFERENCES

Clopper CJ, Pearson E. The Use of Confidence or Fiducial Limits Illustrated in the case of the Binomial. *Biometrika*. 1934;26:404-13.

Miettinen, O. S. and Nurminen, M. Comparative analysis of two rates. *Statistics in Medicine*, 1985;4,213-226.